CLINICAL TRIAL: NCT01431274
Title: A Randomised, Double-blind, Parallel Group Study to Assess the Efficacy and Safety of 52 Weeks of Once Daily Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination (2.5 µg / 5 µg; 5 µg / 5 µg) (Delivered by the Respimat® Inhaler) Compared With the Individual Components (2.5 µg and 5 µg Tiotropium, 5 µg Olodaterol) (Delivered by the Respimat® Inhaler) in Patients With Chronic Obstructive Pulmonary Disease (COPD). [TOnado TM 1]
Brief Title: Tiotropium+Olodaterol Fixed Dose Combination (FDC) Versus Tiotropium and Olodaterol in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.5; 2009-010668-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; Tiotropium Bromide; olodaterol

ARMS (5):
- tiotropium+olodaterol low dose FDC (Experimental): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium + olodaterol; Device: Respimat
- tiotropium+olodaterol high dose FDC (Experimental): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium + olodaterol; Device: Respimat
- olodaterol (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: olodaterol; Device: Respimat
- tiotropium low dose (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium; Device: Respimat
- tiotropium high dose (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium; Device: Respimat

INTERVENTIONS:
Drug: tiotropium + olodaterol — fixed dose combination
  Arms: tiotropium+olodaterol low dose FDC
Drug: tiotropium — low dose
  Arms: tiotropium low dose
Drug: olodaterol — one dose only
  Arms: olodaterol
Drug: tiotropium — high dose
  Arms: tiotropium high dose
Drug: tiotropium + olodaterol — fixed dose combination
  Arms: tiotropium+olodaterol high dose FDC
Device: Respimat — Respimat inhaler

SUMMARY:
The overall objective of this study is to assess the efficacy and safety of 52 weeks once daily treatment with orally inhaled tiotropium + olodaterol FDC (delivered by the RESPIMAT Inhaler) compared with the individual components ( tiotropium, olodaterol) (delivered by the RESPIMAT Inhaler) in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of chronic obstructive pulmonary disease.
2. Relatively stable airway obstruction with post FEV1< 80% predicted normal and post FEV1/FVC <70%.
3. Male or female patients, 40 years of age or older.
4. Smoking history of more than 10 pack years.

Exclusion criteria:

1. Significant disease other than COPD
2. Clinically relevant abnormal lab values.
3. History of asthma.
4. Diagnosis of thyrotoxicosis
5. Diagnosis of paroxysmal tachycardia
6. History of myocardial infarction within 1 year of screening visit
7. Unstable or life-threatening cardiac arrhythmia.
8. Hospitalization for heart failure within the past year.
9. Known active tuberculosis.
10. Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
11. History of life-threatening pulmonary obstruction.
12. History of cystic fibrosis.
13. Clinically evident bronchiectasis.
14. History of significant alcohol or drug abuse.
15. Thoracotomy with pulmonary resection
16. Oral ß-adrenergics.
17. Oral corticosteroid medication at unstable doses
18. Regular use of daytime oxygen therapy for more than one hour per day
19. Pulmonary rehabilitation program in the six weeks prior to the screening visit
20. Investigational drug within one month or six half lives (whichever is greater) prior to screening visit
21. Known hypersensitivity to ß-adrenergic drugs, anticholinergics, BAC, EDTA
22. Pregnant or nursing women.
23. Women of childbearing potential not using a highly effective method of birth control
24. Patients who are unable to comply with pulmonary medication restrictions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2624 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (239):
- United States (35):
  - 1237.5.01038 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1237.5.01036 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1237.5.01015 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 1237.5.01024 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1237.5.01034 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1237.5.01003 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1237.5.01010 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1237.5.01027 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 1237.5.01031 Boehringer Ingelheim Investigational Site, O'Fallon, Illinois
  - 1237.5.01035 Boehringer Ingelheim Investigational Site, Opelousas, Louisiana
  - 1237.5.01004 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1237.5.01017 Boehringer Ingelheim Investigational Site, Biddeford, Maine
  - 1237.5.01028 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1237.5.01013 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 1237.5.01019 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1237.5.01025 Boehringer Ingelheim Investigational Site, Larchmont, New York
  - 1237.5.01008 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1237.5.01023 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1237.5.01016 Boehringer Ingelheim Investigational Site, Tabor City, North Carolina
  - 1237.5.01006 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1237.5.01040 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1237.5.01039 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1237.5.01037 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1237.5.01009 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1237.5.01032 Boehringer Ingelheim Investigational Site, Charleston, Pennsylvania
  - 1237.5.01005 Boehringer Ingelheim Investigational Site, Johnston, Rhode Island
  - 1237.5.01021 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1237.5.01012 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 1237.5.01014 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.5.01029 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1237.5.01002 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1237.5.01026 Boehringer Ingelheim Investigational Site, Lynchburg, Virginia
  - 1237.5.01007 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1237.5.01033 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1237.5.01001 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
- Argentina (13):
  - 1237.5.54010 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1237.5.54013 Boehringer Ingelheim Investigational Site, Caba
  - 1237.5.54016 Boehringer Ingelheim Investigational Site, Caba
  - 1237.5.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1237.5.54002 Boehringer Ingelheim Investigational Site, Cuidad Autonoma de Buenos Airess A
  - 1237.5.54006 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1237.5.54007 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1237.5.54009 Boehringer Ingelheim Investigational Site, Mendoza
  - 1237.5.54012 Boehringer Ingelheim Investigational Site, Monte Grande
  - 1237.5.54008 Boehringer Ingelheim Investigational Site, Quilmes
  - 1237.5.54005 Boehringer Ingelheim Investigational Site, Rosario
  - 1237.5.54004 Boehringer Ingelheim Investigational Site, San Miguel de Tucuma
  - 1237.5.54011 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
- Australia (3):
  - 1237.5.61001 Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - 1237.5.61002 Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - 1237.5.61004 Boehringer Ingelheim Investigational Site, Frankston, Victoria
- Bulgaria (7):
  - 1237.5.35905 Boehringer Ingelheim Investigational Site, Plovdiv
  - 1237.5.35901 Boehringer Ingelheim Investigational Site, Rousse
  - 1237.5.35906 Boehringer Ingelheim Investigational Site, Shumen
  - 1237.5.35902 Boehringer Ingelheim Investigational Site, Sofia
  - 1237.5.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 1237.5.35903 Boehringer Ingelheim Investigational Site, Troyan Municipality
  - 1237.5.35908 Boehringer Ingelheim Investigational Site, Veliko Tarnovo
- Canada (10):
  - 1237.5.02002 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1237.5.02001 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1237.5.02004 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1237.5.02005 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 1237.5.02007 Boehringer Ingelheim Investigational Site, Grimsby, Ontario
  - 1237.5.02011 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1237.5.02003 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1237.5.02006 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1237.5.02008 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1237.5.02009 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (16):
  - 1237.5.86003 Boehringer Ingelheim Investigational Site, Beijing
  - 1237.5.86004 Boehringer Ingelheim Investigational Site, Beijing
  - 1237.5.86011 Boehringer Ingelheim Investigational Site, Changsha
  - 1237.5.86012 Boehringer Ingelheim Investigational Site, Changsha
  - 1237.5.86014 Boehringer Ingelheim Investigational Site, Foshan
  - 1237.5.86001 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1237.5.86015 Boehringer Ingelheim Investigational Site, Nanning
  - 1237.5.86002 Boehringer Ingelheim Investigational Site, Shanghai
  - 1237.5.86005 Boehringer Ingelheim Investigational Site, Shanghai
  - 1237.5.86006 Boehringer Ingelheim Investigational Site, Shanghai
  - 1237.5.86007 Boehringer Ingelheim Investigational Site, Shanghai
  - 1237.5.86009 Boehringer Ingelheim Investigational Site, Shenyang
  - 1237.5.86016 Boehringer Ingelheim Investigational Site, Wuhan
  - 1237.5.86010 Boehringer Ingelheim Investigational Site, Xi'an
  - 1237.5.86008 Boehringer Ingelheim Investigational Site, Yangzhou
  - 1237.5.86017 Boehringer Ingelheim Investigational Site, Yinchuan
- Czechia (5):
  - 1237.5.42004 Boehringer Ingelheim Investigational Site, Beroun
  - 1237.5.42002 Boehringer Ingelheim Investigational Site, Cvikov
  - 1237.5.42001 Boehringer Ingelheim Investigational Site, Prague
  - 1237.5.42005 Boehringer Ingelheim Investigational Site, Rokycany
  - 1237.5.42003 Boehringer Ingelheim Investigational Site, Znojmo
- Denmark (10):
  - 1237.5.45002 Boehringer Ingelheim Investigational Site, Aalborg
  - 1237.5.45009 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1237.5.45007 Boehringer Ingelheim Investigational Site, Kolding
  - 1237.5.45001 Boehringer Ingelheim Investigational Site, København NV
  - 1237.5.45011 Boehringer Ingelheim Investigational Site, Næstved
  - 1237.5.45006 Boehringer Ingelheim Investigational Site, Odense C
  - 1237.5.45008 Boehringer Ingelheim Investigational Site, Roskilde
  - 1237.5.45003 Boehringer Ingelheim Investigational Site, Silkeborg
  - 1237.5.45005 Boehringer Ingelheim Investigational Site, Sønderborg
  - 1237.5.45004 Boehringer Ingelheim Investigational Site, Vaerløse
- Estonia (2):
  - 1237.5.37002 Boehringer Ingelheim Investigational Site, Tallinn
  - 1237.5.37001 Boehringer Ingelheim Investigational Site, Tartu
- Finland (3):
  - 1237.5.35801 Boehringer Ingelheim Investigational Site, Helsinki
  - 1237.5.35804 Boehringer Ingelheim Investigational Site, Pori
  - 1237.5.35802 Boehringer Ingelheim Investigational Site, Turku
- France (7):
  - 1237.5.33004 Boehringer Ingelheim Investigational Site, Béthune
  - 1237.5.33007 Boehringer Ingelheim Investigational Site, Montpellier
  - 1237.5.33005 Boehringer Ingelheim Investigational Site, Nantes
  - 1237.5.33006 Boehringer Ingelheim Investigational Site, Nîmes
  - 1237.5.33008 Boehringer Ingelheim Investigational Site, Perpignan
  - 1237.5.33001 Boehringer Ingelheim Investigational Site, Saint-Pierre
  - 1237.5.33002 Boehringer Ingelheim Investigational Site, Strasbourg
- Germany (13):
  - 1237.5.49006 Boehringer Ingelheim Investigational Site, Bamberg
  - 1237.5.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.5.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.5.49013 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.5.49011 Boehringer Ingelheim Investigational Site, Erfurt
  - 1237.5.49005 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.5.49010 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.5.49009 Boehringer Ingelheim Investigational Site, Koblenz
  - 1237.5.49014 Boehringer Ingelheim Investigational Site, Neu-Isenburg
  - 1237.5.49012 Boehringer Ingelheim Investigational Site, Oschersleben
  - 1237.5.49001 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1237.5.49004 Boehringer Ingelheim Investigational Site, Weinheim
  - 1237.5.49008 Boehringer Ingelheim Investigational Site, Wiesloch
- Guatemala (7):
  - 1237.5.50201 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.5.50202 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.5.50203 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.5.50204 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.5.50205 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.5.50206 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.5.50207 Boehringer Ingelheim Investigational Site, Guatemala City
- Hungary (5):
  - 1237.5.36005 Boehringer Ingelheim Investigational Site, Debrecen
  - 1237.5.36001 Boehringer Ingelheim Investigational Site, Deszk
  - 1237.5.36006 Boehringer Ingelheim Investigational Site, Kapuvár
  - 1237.5.36003 Boehringer Ingelheim Investigational Site, Szombathely
  - 1237.5.36002 Boehringer Ingelheim Investigational Site, Törökbálint
- India (9):
  - 1237.5.91010 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1237.5.91002 Boehringer Ingelheim Investigational Site, Bangalore
  - 1237.5.91007 Boehringer Ingelheim Investigational Site, Bangalore
  - 1237.5.91004 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1237.5.91011 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1237.5.91001 Boehringer Ingelheim Investigational Site, Jaipur
  - 1237.5.91008 Boehringer Ingelheim Investigational Site, Jaipur
  - 1237.5.91009 Boehringer Ingelheim Investigational Site, Mysore
  - 1237.5.91006 Boehringer Ingelheim Investigational Site, Pune
- Italy (6):
  - 1237.5.39008 Boehringer Ingelheim Investigational Site, Cagliari
  - 1237.5.39002 Boehringer Ingelheim Investigational Site, Genova
  - 1237.5.39006 Boehringer Ingelheim Investigational Site, Montescano (PV)
  - 1237.5.39009 Boehringer Ingelheim Investigational Site, Monza
  - 1237.5.39004 Boehringer Ingelheim Investigational Site, Parma
  - 1237.5.39001 Boehringer Ingelheim Investigational Site, Pisa
- Japan (45):
  - 1237.5.81003 Boehringer Ingelheim Investigational Site, Aoba-ku, Sendai, Miyagi
  - 1237.5.81001 Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - 1237.5.81006 Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - 1237.5.81044 Boehringer Ingelheim Investigational Site, Chuo-ku, Kumamoto, Kumamoto
  - 1237.5.81035 Boehringer Ingelheim Investigational Site, Gifu, Gifu
  - 1237.5.81017 Boehringer Ingelheim Investigational Site, Hakata-ku, Fukuoka, Fukuoka
  - 1237.5.81031 Boehringer Ingelheim Investigational Site, Hamamatsushi, Shizuoka
  - 1237.5.81014 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1237.5.81037 Boehringer Ingelheim Investigational Site, Ikoma, Nara
  - 1237.5.81024 Boehringer Ingelheim Investigational Site, Inashiki-gun, Ibaraki
  - 1237.5.81008 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 1237.5.81016 Boehringer Ingelheim Investigational Site, Jonan-ku, Fukuoka, Fukuoka
  - 1237.5.81020 Boehringer Ingelheim Investigational Site, Kagoshima, Kagoshima,
  - 1237.5.81021 Boehringer Ingelheim Investigational Site, Kagoshima, Kagoshima
  - 1237.5.81005 Boehringer Ingelheim Investigational Site, Kamogawa, Chiba
  - 1237.5.81011 Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - 1237.5.81018 Boehringer Ingelheim Investigational Site, Kitakyusyu,Fukuoka
  - 1237.5.81042 Boehringer Ingelheim Investigational Site, Koga, Fukuoka
  - 1237.5.81032 Boehringer Ingelheim Investigational Site, Komaki, Aichi
  - 1237.5.81033 Boehringer Ingelheim Investigational Site, Komaki, Aichi
  - 1237.5.81019 Boehringer Ingelheim Investigational Site, Koshi, Kumamoto
  - 1237.5.81027 Boehringer Ingelheim Investigational Site, Koto-ku, Tokyo
  - 1237.5.81025 Boehringer Ingelheim Investigational Site, Kuki, Saitama
  - 1237.5.81038 Boehringer Ingelheim Investigational Site, Kure, Hiroshima
  - 1237.5.81015 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 1237.5.81029 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1237.5.81030 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1237.5.81010 Boehringer Ingelheim Investigational Site, Matsusaka, Mie
  - 1237.5.81041 Boehringer Ingelheim Investigational Site, Minami-ku. Fukuoka, Fukuoka
  - 1237.5.81002 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 1237.5.81034 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1237.5.81036 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1237.5.81004 Boehringer Ingelheim Investigational Site, Naka-gun, Ibaraki
  - 1237.5.81022 Boehringer Ingelheim Investigational Site, Okinawa, Urasoe
  - 1237.5.81023 Boehringer Ingelheim Investigational Site, Okinawa, Urasoe
  - 1237.5.81012 Boehringer Ingelheim Investigational Site, Sayama, Osaka
  - 1237.5.81045 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1237.5.81009 Boehringer Ingelheim Investigational Site, Seto, Aichi
  - 1237.5.81026 Boehringer Ingelheim Investigational Site, Shinagawa, Tokyo
  - 1237.5.81007 Boehringer Ingelheim Investigational Site, Shinjyuku-ku, Tokyo
  - 1237.5.81039 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
  - 1237.5.81040 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
  - 1237.5.81013 Boehringer Ingelheim Investigational Site, Wakayama, Wakayama
  - 1237.5.81043 Boehringer Ingelheim Investigational Site, Yanagawa-shi, Fukuoka,
  - 1237.5.81028 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
- Mexico (4):
  - 1237.5.52002 Boehringer Ingelheim Investigational Site, Hermosillo
  - 1237.5.52003 Boehringer Ingelheim Investigational Site, México
  - 1237.5.52007 Boehringer Ingelheim Investigational Site, Monterrey
  - 1237.5.52001 Boehringer Ingelheim Investigational Site, Tijuana
- Netherlands (10):
  - 1237.5.31004 Boehringer Ingelheim Investigational Site, Almelo
  - 1237.5.31006 Boehringer Ingelheim Investigational Site, Breda
  - 1237.5.31001 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1237.5.31008 Boehringer Ingelheim Investigational Site, Harderwijk
  - 1237.5.31007 Boehringer Ingelheim Investigational Site, Heerlen
  - 1237.5.31010 Boehringer Ingelheim Investigational Site, Hengelo
  - 1237.5.31009 Boehringer Ingelheim Investigational Site, Hoorn
  - 1237.5.31005 Boehringer Ingelheim Investigational Site, Nieuwegein
  - 1237.5.31002 Boehringer Ingelheim Investigational Site, Veldhoven
  - 1237.5.31003 Boehringer Ingelheim Investigational Site, Zutphen
- New Zealand (2):
  - 1237.5.64002 Boehringer Ingelheim Investigational Site, Dunedin
  - 1237.5.64001 Boehringer Ingelheim Investigational Site, Greenlane East Auckland NZ
- Portugal (7):
  - 1237.5.35105 Boehringer Ingelheim Investigational Site, Amadora
  - 1237.5.35101 Boehringer Ingelheim Investigational Site, Coimbra
  - 1237.5.35102 Boehringer Ingelheim Investigational Site, Lisbon
  - 1237.5.35104 Boehringer Ingelheim Investigational Site, Lisbon
  - 1237.5.35103 Boehringer Ingelheim Investigational Site, Porto
  - 1237.5.35106 Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
  - 1237.5.35107 Boehringer Ingelheim Investigational Site, Viseu
- Russia (5):
  - 1237.5.07001 Boehringer Ingelheim Investigational Site, Gatchina (Leningradskaya Oblast)
  - 1237.5.07003 Boehringer Ingelheim Investigational Site, Kazan'
  - 1237.5.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.5.07005 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.5.07002 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovenia (2):
  - 1237.5.38601 Boehringer Ingelheim Investigational Site, Golnik
  - 1237.5.38602 Boehringer Ingelheim Investigational Site, Golnik
- South Korea (8):
  - 1237.5.82004 Boehringer Ingelheim Investigational Site, Bucheon-si
  - 1237.5.82008 Boehringer Ingelheim Investigational Site, Daegu
  - 1237.5.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.5.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.5.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.5.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.5.82005 Boehringer Ingelheim Investigational Site, Suwon
  - 1237.5.82006 Boehringer Ingelheim Investigational Site, Wŏnju
- Turkey (Türkiye) (5):
  - 1237.5.90003 Boehringer Ingelheim Investigational Site, Istanbul
  - 1237.5.90004 Boehringer Ingelheim Investigational Site, Istanbul
  - 1237.5.90002 Boehringer Ingelheim Investigational Site, Izmir
  - 1237.5.90005 Boehringer Ingelheim Investigational Site, İzmit
  - 1237.5.90001 Boehringer Ingelheim Investigational Site, Mersin

REFERENCES:
- [Derived] Rabe KF, Chalmers JD, Miravitlles M, Kocks JWH, Tsiligianni I, de la Hoz A, Xue W, Singh D, Ferguson GT, Wedzicha J. Tiotropium/Olodaterol Delays Clinically Important Deterioration Compared with Tiotropium Monotherapy in Patients with Early COPD: a Post Hoc Analysis of the TONADO(R) Trials. Adv Ther. 2021 Jan;38(1):579-593. doi: 10.1007/s12325-020-01528-2. Epub 2020 Nov 11. PMID 33175291
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Andreas S, Bothner U, de la Hoz A, Kloer I, Trampisch M, Alter P. No Influence on Cardiac Arrhythmia or Heart Rate from Long-Term Treatment with Tiotropium/Olodaterol versus Monocomponents by Holter ECG Analysis in Patients with Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1945-1953. doi: 10.2147/COPD.S246350. eCollection 2020. PMID 32848380
- [Derived] Andreas S, McGarvey L, Bothner U, Trampisch M, de la Hoz A, Flezar M, Buhl R, Alter P. Absence of Adverse Effects of Tiotropium/Olodaterol Compared with the Monocomponents on Long-Term Heart Rate and Blood Pressure in Patients with Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1935-1944. doi: 10.2147/COPD.S246348. eCollection 2020. PMID 32848379
- [Derived] Wedzicha JA, Buhl R, Singh D, Vogelmeier CF, de la Hoz A, Xue W, Anzueto A, Calverley PMA. Tiotropium/Olodaterol Decreases Exacerbation Rates Compared with Tiotropium in a Range of Patients with COPD: Pooled Analysis of the TONADO(R)/DYNAGITO(R) Trials. Adv Ther. 2020 Oct;37(10):4266-4279. doi: 10.1007/s12325-020-01438-3. Epub 2020 Aug 10. PMID 32776202
- [Derived] Buhl R, de la Hoz A, Xue W, Singh D, Ferguson GT. Efficacy of Tiotropium/Olodaterol Compared with Tiotropium as a First-Line Maintenance Treatment in Patients with COPD Who Are Naive to LAMA, LABA and ICS: Pooled Analysis of Four Clinical Trials. Adv Ther. 2020 Oct;37(10):4175-4189. doi: 10.1007/s12325-020-01411-0. Epub 2020 Jul 15. PMID 32671684
- [Derived] Buhl R, Singh D, de la Hoz A, Xue W, Ferguson GT. Benefits of Tiotropium/Olodaterol Compared with Tiotropium in Patients with COPD Receiving only LAMA at Baseline: Pooled Analysis of the TONADO(R) and OTEMTO(R) Studies. Adv Ther. 2020 Aug;37(8):3485-3499. doi: 10.1007/s12325-020-01373-3. Epub 2020 May 27. PMID 32462607
- [Derived] Ferguson GT, Buhl R, Bothner U, Hoz A, Voss F, Anzueto A, Calverley PMA. Safety of tiotropium/olodaterol in chronic obstructive pulmonary disease: pooled analysis of three large, 52-week, randomized clinical trials. Respir Med. 2018 Oct;143:67-73. doi: 10.1016/j.rmed.2018.08.012. Epub 2018 Aug 28. PMID 30261995
- [Derived] Maltais F, Buhl R, Koch A, Amatto VC, Reid J, Gronke L, Bothner U, Voss F, McGarvey L, Ferguson GT. beta-Blockers in COPD: A Cohort Study From the TONADO Research Program. Chest. 2018 Jun;153(6):1315-1325. doi: 10.1016/j.chest.2018.01.008. Epub 2018 Jan 31. PMID 29355547
- [Derived] Buhl R, Magder S, Bothner U, Tetzlaff K, Voss F, Loaiza L, Vogelmeier CF, McGarvey L. Long-term general and cardiovascular safety of tiotropium/olodaterol in patients with moderate to very severe chronic obstructive pulmonary disease. Respir Med. 2017 Jan;122:58-66. doi: 10.1016/j.rmed.2016.11.011. Epub 2016 Nov 14. PMID 27993292
- [Derived] Ferguson GT, Flezar M, Korn S, Korducki L, Gronke L, Abrahams R, Buhl R. Efficacy of Tiotropium + Olodaterol in Patients with Chronic Obstructive Pulmonary Disease by Initial Disease Severity and Treatment Intensity: A Post Hoc Analysis. Adv Ther. 2015 Jun;32(6):523-36. doi: 10.1007/s12325-015-0218-0. Epub 2015 Jun 26. PMID 26112656
- [Derived] Buhl R, Maltais F, Abrahams R, Bjermer L, Derom E, Ferguson G, Flezar M, Hebert J, McGarvey L, Pizzichini E, Reid J, Veale A, Gronke L, Hamilton A, Korducki L, Tetzlaff K, Waitere-Wijker S, Watz H, Bateman E. Tiotropium and olodaterol fixed-dose combination versus mono-components in COPD (GOLD 2-4). Eur Respir J. 2015 Apr;45(4):969-79. doi: 10.1183/09031936.00136014. Epub 2015 Jan 8. PMID 25573406

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial was one of 2 confirmatory Phase III 52-week, multi-centre, multi-national, randomised,double-blind, parallel group studies to evaluate the long-term efficacy and safety of once daily treatment with orally inhaled Tio+Olo FDC (2.5/5μg; 5/5μg) compared with the individual components (2.5μg; 5μg Tiotropium, 5μg Olodaterol) in COPD patients
Groups:
- Olodaterol (5 μg): Oral inhalation of Olodaterol 5 μg (2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tiotropium (2.5 μg): Oral inhalation of Tiotropium 2.5 μg (1.25 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tiotropium (5 μg): Oral inhalation of Tiotropium 5 μg (2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo FDC (2.5/5 μg): Oral inhalation of fixed dose combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg (Tiotropium: 1.25 μg per actuation and Olodaterol: 2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo FDC (5/5 μg): Oral inhalation of FDC of Tiotropium 5 μg and Olodaterol 5 μg (Tiotropium and Olodaterol: 2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
Period: Overall Study
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Started | 528 | 525 | 527 | 522 | 522
Completed | 431 | 448 | 455 | 462 | 466
Not Completed | 97 | 77 | 72 | 60 | 56
Not completed — Adverse Event | 51 | 37 | 43 | 30 | 37
Not completed — Consent withdrawn not due to AE | 29 | 20 | 17 | 20 | 11
Not completed — Non compliant with protocol | 5 | 8 | 4 | 4 | 4
Not completed — Lost to Follow-up | 6 | 7 | 1 | 4 | 0
Not completed — Other reason not stated above | 6 | 5 | 7 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all patients in the randomised set who were dispensed study medication and were documented to have taken any dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg) | Total
Number analyzed (Participants) | 528 | 525 | 527 | 522 | 522 | 2624
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.0) | 64.2 (8.6) | 64.2 (8.5) | 64.1 (8.0) | 64.8 (8.2) | 64.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 133 | 144 | 133 | 138 | 690
  Male | 386 | 392 | 383 | 389 | 384 | 1934

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) (0-3h) Response on Day 169.
Description: FEV1 AUC(0-3h) was calculated as the area under the FEV1- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres. FEV1 AUC(0-3h) response was defined as FEV1 AUC(0-3h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom. Number of participants analyzed are the number of patients contributing to the MMRM model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 169 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on Day 169.
Population: The Full analysis set (FAS) included all patients who were randomised, who were dispensed study medication, were documented to have taken any dose of study medication and who had a non-missing baseline and at least one non-missing post-baseline measurement before or at Week 24 for any of the primary and key secondary efficacy endpoints.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.133 (0.008) | 0.148 (0.008) | 0.139 (0.008) | 0.241 (0.008) | 0.256 (0.008)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.123, 95% CI 2-sided [0.100 to 0.146], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.117, 95% CI [0.094 to 0.140], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.109, 95% CI 2-sided [0.086 to 0.132], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.093, 95% CI 2-sided [0.070 to 0.116], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.102, 95% CI 2-sided [0.080 to 0.125], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2169, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.014, 95% CI 2-sided [-0.008 to 0.037], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.108, 95% CI 2-sided [0.085 to 0.130], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.5849, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.006, 95% CI 2-sided [-0.017 to 0.029], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1863, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.016, 95% CI 2-sided [-0.007 to 0.039], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4352, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.009, 95% CI 2-sided [-0.032 to 0.014], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

2. Primary Outcome: Trough FEV1 Response on Day 170.
Description: Trough FEV1 was defined as the FEV1 value at the end of the dosing interval (24 hours) and was calculated as the mean of the 2 FEV1 measurements performed at 23 h and at 23 h 50 min after inhalation of study medication at the clinic visit on the previous day.
  Trough FEV1 response was defined as trough FEV1 minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an MMRM including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 23 h and at 23 h 50 min after inhalation of study medication on Day 170
Population: FAS. Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.054 (0.009) | 0.083 (0.008) | 0.065 (0.008) | 0.111 (0.008) | 0.136 (0.008)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.082, 95% CI 2-sided [0.059 to 0.106], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.071, 95% CI 2-sided [0.047 to 0.094], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.058, 95% CI 2-sided [0.034 to 0.081], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0174, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.029, 95% CI 2-sided [0.005 to 0.052], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.046, 95% CI 2-sided [0.023 to 0.070], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0407, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.024, 95% CI 2-sided [0.001 to 0.048], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Mean Difference (Final Values) = 0.053, 95% CI 2-sided [0.030 to 0.077], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.3326, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.012, 95% CI 2-sided [-0.012 to 0.035], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0151, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.029, 95% CI 2-sided [0.006 to 0.053], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1421, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.018, 95% CI 2-sided [-0.041 to 0.006], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

3. Primary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score on Day 169 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: The SGRQ is designed to measure health impairment in patients with COPD. It is divided into 2 parts: part 1 produces the symptoms score, and part 2 the activity and impacts scores. A total score is also produced. Each subscale score is the sum of the weights for the items in the subscale as a percent of the sum of the weights for a patient in the worst possible condition. The total score uses the same calculation except that the weights are summed over the entire questionnaire. The individual subscales as well as the total score can range from 0 to 100 with a lower score denoting a better health status. Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 169
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 954 | 960 | 954 | 990 | 979
points on a scale | 38.366 (0.396) | 37.792 (0.390) | 37.907 (0.393) | 37.335 (0.385) | 36.674 (0.386)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.693, 95% CI 2-sided [-2.778 to -0.608], Standard Error of Mean 0.553 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0252, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.233, 95% CI 2-sided [-2.313 to -0.153], Standard Error of Mean 0.551 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0620, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.031, 95% CI 2-sided [-2.113 to 0.052], Standard Error of Mean 0.552 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.4051, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.456, 95% CI 2-sided [-1.531 to 0.618], Standard Error of Mean 0.548 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.2988, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.571, 95% CI 2-sided [-1.649 to 0.507], Standard Error of Mean 0.550 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2249, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.662, 95% CI 2-sided [-1.731 to 0.407], Standard Error of Mean 0.545 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0418, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.118, 95% CI 2-sided [-2.195 to -0.042], Standard Error of Mean 0.549 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4097, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.460, 95% CI 2-sided [-1.552 to 0.633], Standard Error of Mean 0.557 — Tiotropium (2.5 µg) versus Olodaterol (5 µg) Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.3013, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.575, 95% CI 2-sided [-1.664 to 0.515], Standard Error of Mean 0.556 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8355, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.115, 95% CI 2-sided [-0.970 to 1.200], Standard Error of Mean 0.554 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors

4. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 169 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: Mahler Transitional Dyspnoea Index (TDI) focal score on Day 169 From the Two Twin Trials, present 1237.5 (NCT01431274) and 1237.6 (NCT01431287) is the key secondary endpoint.
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome. Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 169
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.564 (0.096) | 1.690 (0.095) | 1.627 (0.096) | 1.980 (0.095) | 1.983 (0.095)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.420, 95% CI 2-sided [0.155 to 0.684], Standard Error of Mean 0.135 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0082, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.356, 95% CI 2-sided [0.092 to 0.619], Standard Error of Mean 0.135 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.416, 95% CI 2-sided [0.152 to 0.681], Standard Error of Mean 0.135 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0307, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.290, 95% CI 2-sided [0.027 to 0.554], Standard Error of Mean 0.134 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0088, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.352, 95% CI 2-sided [0.089 to 0.616], Standard Error of Mean 0.135 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.9801, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.003, 95% CI 2-sided [-0.259 to 0.266], Standard Error of Mean 0.134 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0289, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.294, 95% CI 2-sided [0.030 to 0.557], Standard Error of Mean 0.134 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6382, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.064, 95% CI 2-sided [-0.202 to 0.330], Standard Error of Mean 0.136 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.3525, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.126, 95% CI 2-sided [-0.140 to 0.391], Standard Error of Mean 0.135 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6457, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.062, 95% CI 2-sided [-0.327 to 0.203], Standard Error of Mean 0.135 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

5. Secondary Outcome: FEV1 AUC(0-3h) Response on Day 1
Description: FEV1 AUC(0-3h) was calculated as the area under the FEV1- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres.
  FEV1 AUC(0-3h) response was defined as FEV1 AUC(0-3h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose of randomised treatment at Day1.
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on the first day of randomized treatment.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.205 (0.009) | 0.148 (0.009) | 0.157 (0.009) | 0.226 (0.009) | 0.237 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0067, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.033, 95% CI 2-sided [0.009 to 0.056], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.081, 95% CI 2-sided [0.057 to 0.104], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0746, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.022, 95% CI 2-sided [-0.002 to 0.045], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.078, 95% CI 2-sided [0.054 to 0.101], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.070, 95% CI 2-sided [0.046 to 0.093], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.3549, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.011, 95% CI 2-sided [-0.013 to 0.035], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.089, 95% CI 2-sided [0.065 to 0.113], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.048, 95% CI 2-sided [-0.072 to -0.025], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.056, 95% CI 2-sided [-0.080 to -0.033], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.5018, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.008, 95% CI 2-sided [-0.016 to 0.032], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

6. Secondary Outcome: FEV1 AUC(0-3h) Response on Day 85
Description: as for outcome 5
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 85 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on Day 85.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.161 (0.009) | 0.176 (0.009) | 0.162 (0.009) | 0.271 (0.009) | 0.289 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.128, 95% CI 2-sided [0.104 to 0.152], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.126, 95% CI 2-sided [0.102 to 0.150], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.111, 95% CI 2-sided [0.087 to 0.135], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.096, 95% CI 2-sided [0.072 to 0.120], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.109, 95% CI 2-sided [0.085 to 0.133], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1569, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.017, 95% CI 2-sided [-0.007 to 0.041], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.113, 95% CI 2-sided [0.089 to 0.137], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8834, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.002, 95% CI 2-sided [-0.022 to 0.026], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2129, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.015, 95% CI 2-sided [-0.009 to 0.039], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.2702, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.013, 95% CI 2-sided [-0.037 to 0.010], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

7. Secondary Outcome: FEV1 AUC(0-3h) Response on Day 365
Description: as for outcome 5
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 365 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on Day 365.
Population: FAS (on day 365). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.096 (0.009) | 0.116 (0.009) | 0.122 (0.009) | 0.214 (0.009) | 0.237 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.141, 95% CI 2-sided [0.117 to 0.166], Standard Error of Mean 0.013 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.115, 95% CI 2-sided [0.090 to 0.139], Standard Error of Mean 0.013 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.119, 95% CI 2-sided [0.094 to 0.143], Standard Error of Mean 0.013 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.099, 95% CI 2-sided [0.074 to 0.123], Standard Error of Mean 0.013 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.092, 95% CI 2-sided [0.067 to 0.117], Standard Error of Mean 0.013 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0717, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.023, 95% CI 2-sided [-0.002 to 0.047], Standard Error of Mean 0.013 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.121, 95% CI 2-sided [0.097 to 0.146], Standard Error of Mean 0.013 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0344, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.027, 95% CI 2-sided [0.002 to 0.051], Standard Error of Mean 0.013 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1126, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.020, 95% CI 2-sided [-0.005 to 0.045], Standard Error of Mean 0.013 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6009, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.007, 95% CI 2-sided [-0.018 to 0.031], Standard Error of Mean 0.013 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

8. Secondary Outcome: Trough FEV1 Response on Day 15.
Description: Trough FEV1 was defined as the FEV1 value at the end of the dosing interval (24 hours), calculated as the mean of the pre-dose measurements.
  Trough FEV1 response was defined as trough FEV1 minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed
  1 h and 10 min prior to administration of the first dose of randomised treatment at Day1.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 15
Population: FAS (day 15). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.085 (0.009) | 0.101 (0.009) | 0.094 (0.009) | 0.132 (0.009) | 0.157 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.072, 95% CI 2-sided [0.049 to 0.096], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.063, 95% CI 2-sided [0.039 to 0.087], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.047, 95% CI 2-sided [0.023 to 0.070], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0122, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.030, 95% CI 2-sided [0.007 to 0.054], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.037, 95% CI 2-sided [0.014 to 0.061], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0347, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.026, 95% CI 2-sided [0.002 to 0.049], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.056, 95% CI 2-sided [0.032 to 0.080], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4407, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.009, 95% CI 2-sided [-0.014 to 0.033], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1777, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.016, 95% CI 2-sided [-0.007 to 0.040], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.5641, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.007, 95% CI 2-sided [-0.031 to 0.017], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

9. Secondary Outcome: Trough FEV1 Response on Day 43
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 43.
Population: FAS (day 43). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.083 (0.009) | 0.097 (0.009) | 0.088 (0.009) | 0.120 (0.009) | 0.163 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.080, 95% CI 2-sided [0.057 to 0.104], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.075, 95% CI 2-sided [0.051 to 0.099], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.038, 95% CI 2-sided [0.014 to 0.062], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0517, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.024, 95% CI 2-sided [-0.000 to 0.047], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0072, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.033, 95% CI 2-sided [0.009 to 0.056], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.042, 95% CI 2-sided [0.019 to 0.066], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.066, 95% CI 2-sided [0.042 to 0.090], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6619, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.005, 95% CI 2-sided [-0.018 to 0.029], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2401, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.014, 95% CI 2-sided [-0.010 to 0.038], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4601, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.009, 95% CI 2-sided [-0.033 to 0.015], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

10. Secondary Outcome: Trough FEV1 Response on Day 85
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 1 hr and 10 min pre-dose on day 85.
Population: FAS (day 85). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.057 (0.009) | 0.077 (0.009) | 0.070 (0.009) | 0.128 (0.009) | 0.146 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.088, 95% CI 2-sided [0.064 to 0.112], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.076, 95% CI 2-sided [0.052 to 0.100], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.070, 95% CI 2-sided [0.046 to 0.094], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.051, 95% CI 2-sided [0.027 to 0.075], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.058, 95% CI 2-sided [0.034 to 0.082], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1405, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.018, 95% CI 2-sided [-0.006 to 0.042], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.069, 95% CI 2-sided [0.045 to 0.093], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.3118, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.012, 95% CI 2-sided [-0.012 to 0.036], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1171, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.019, 95% CI 2-sided [-0.005 to 0.043], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.5759, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.007, 95% CI 2-sided [-0.031 to 0.017], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

11. Secondary Outcome: Trough FEV1 Response on Day 169
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 1 hr and 10 min pre-dose on Day 169
Population: FAS (day 169). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.033 (0.009) | 0.047 (0.009) | 0.050 (0.009) | 0.094 (0.009) | 0.112 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.079, 95% CI 2-sided [0.055 to 0.103], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.062, 95% CI 2-sided [0.038 to 0.086], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.061, 95% CI 2-sided [0.037 to 0.085], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.047, 95% CI 2-sided [0.022 to 0.071], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.044, 95% CI 2-sided [0.019 to 0.068], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1360, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.018, 95% CI 2-sided [-0.006 to 0.042], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.065, 95% CI 2-sided [0.041 to 0.089], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1617, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.017, 95% CI 2-sided [-0.007 to 0.041], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2476, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.014, 95% CI 2-sided [-0.010 to 0.039], Standard Error of Mean 0.012 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8083, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.003, 95% CI 2-sided [-0.021 to 0.027], Standard Error of Mean 0.012 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

12. Secondary Outcome: Trough FEV1 Response on Day 365
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 1 hr and 10 min pre-dose on day 365
Population: FAS (day 365). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | -0.000 (0.009) | 0.028 (0.009) | 0.036 (0.009) | 0.075 (0.009) | 0.099 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.100, 95% CI 2-sided [0.075 to 0.124], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.064, 95% CI 2-sided [0.039 to 0.088], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.076, 95% CI 2-sided [0.051 to 0.100], Standard Error of Mean 0.013 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.048, 95% CI 2-sided [0.023 to 0.072], Standard Error of Mean 0.013 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.040, 95% CI 2-sided [0.015 to 0.064], Standard Error of Mean 0.012 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0554, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.024, 95% CI 2-sided [-0.001 to 0.048], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.071, 95% CI 2-sided [0.047 to 0.096], Standard Error of Mean 0.012 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.036, 95% CI 2-sided [0.011 to 0.060], Standard Error of Mean 0.013 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0248, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.028, 95% CI 2-sided [0.004 to 0.053], Standard Error of Mean 0.013 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.5338, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.008, 95% CI 2-sided [-0.017 to 0.032], Standard Error of Mean 0.013 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

13. Secondary Outcome: FVC (Forced Vital Capacity) AUC(0-3h) Response on Day 1
Description: FVC AUC(0-3h) was calculated as the area under the FVC- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres.
  FVC AUC(0-3h) response was defined as FVC AUC(0-3h) minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: as for outcome 5
Population: FAS (day 1). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.350 (0.017) | 0.277 (0.017) | 0.289 (0.017) | 0.400 (0.017) | 0.427 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.077, 95% CI 2-sided [0.029 to 0.125], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.138, 95% CI 2-sided [0.090 to 0.186], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0426, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.050, 95% CI 2-sided [0.002 to 0.098], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.122, 95% CI [0.074 to 0.170], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.111, 95% CI 2-sided [0.063 to 0.159], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2661, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.027, 95% CI 2-sided [-0.021 to 0.075], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.150, 95% CI 2-sided [0.102 to 0.198], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0119, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.061, 95% CI 2-sided [-0.109 to -0.014], Standard Error of Mean 0.024 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.073, 95% CI 2-sided [-0.121 to -0.025], Standard Error of Mean 0.024 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6408, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.011, 95% CI 2-sided [-0.036 to 0.059], Standard Error of Mean 0.024 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

14. Secondary Outcome: FVC (Forced Vital Capacity) AUC(0-3h) Response on Day 85
Description: FVC AUC(0-3h) was calculated as the area under the FVC- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres.
  FVC AUC(0-3h) response was defined as FVC AUC(0-3h) minus baseline FVC.Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.247 (0.017) | 0.318 (0.017) | 0.275 (0.017) | 0.432 (0.017) | 0.469 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.221, 95% CI 2-sided [0.173 to 0.270], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.193, 95% CI 2-sided [0.145 to 0.242], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.185, 95% CI 2-sided [0.136 to 0.233], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.114, 95% CI 2-sided [0.065 to 0.162], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.157, 95% CI 2-sided [0.108 to 0.205], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1355, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.037, 95% CI 2-sided [-0.012 to 0.085], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.151, 95% CI 2-sided [0.102 to 0.199], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.2562, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.028, 95% CI 2-sided [-0.020 to 0.076], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.071, 95% CI 2-sided [0.022 to 0.119], Standard Error of Mean 0.025 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0815, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.043, 95% CI 2-sided [-0.091 to 0.005], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

15. Secondary Outcome: FVC (Forced Vital Capacity) AUC(0-3h) Response on Day 169
Description: as for outcome 13
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.212 (0.017) | 0.279 (0.017) | 0.254 (0.017) | 0.386 (0.017) | 0.407 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.195, 95% CI 2-sided [0.149 to 0.242], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.153, 95% CI 2-sided [0.107 to 0.199], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.174, 95% CI 2-sided [0.128 to 0.221], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.107, 95% CI 2-sided [0.061 to 0.154], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.132, 95% CI 2-sided [0.086 to 0.178], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.3727, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.021, 95% CI 2-sided [-0.025 to 0.067], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.128, 95% CI 2-sided [0.082 to 0.175], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0744, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.042, 95% CI 2-sided [-0.004 to 0.089], Standard Error of Mean 0.024 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0047, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.067, 95% CI 2-sided [0.021 to 0.114], Standard Error of Mean 0.024 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.2945, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.025, 95% CI 2-sided [-0.071 to 0.022], Standard Error of Mean 0.024 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

16. Secondary Outcome: FVC (Forced Vital Capacity) AUC(0-3h) Response on Day 365
Description: as for outcome 13
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 525 | 524 | 526 | 521 | 522
Litres | 0.172 (0.018) | 0.241 (0.018) | 0.221 (0.018) | 0.364 (0.018) | 0.377 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.205, 95% CI 2-sided [0.155 to 0.255], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.156, 95% CI 2-sided [0.107 to 0.206], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.192, 95% CI 2-sided [0.142 to 0.242], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.124, 95% CI 2-sided [0.074 to 0.174], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.144, 95% CI 2-sided [0.094 to 0.193], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.6103, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.013, 95% CI 2-sided [-0.037 to 0.062], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.137, 95% CI 2-sided [0.087 to 0.186], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0559, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.049, 95% CI 2-sided [-0.001 to 0.098], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.068, 95% CI 2-sided [0.018 to 0.118], Standard Error of Mean 0.025 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4368, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.020, 95% CI 2-sided [-0.070 to 0.030], Standard Deviation 0.025 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

17. Secondary Outcome: Trough FVC Response on Day 15.
Description: Trough FVC was defined as the FVC value at the end of the dosing interval (24 hours), calculated as the mean of the pre-dose measurements.
  Trough FVC response was defined as trough FVC minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 15
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.149 (0.018) | 0.222 (0.018) | 0.220 (0.018) | 0.270 (0.018) | 0.296 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.147, 95% CI 2-sided [0.098 to 0.196], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.076, 95% CI 2-sided [0.027 to 0.125], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.121, 95% CI 2-sided [0.072 to 0.170], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0545, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.048, 95% CI 2-sided [-0.001 to 0.097], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0456, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.050, 95% CI 2-sided [0.001 to 0.099], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2949, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.026, 95% CI 2-sided [-0.023 to 0.075], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.074, 95% CI 2-sided [0.025 to 0.123], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.071, 95% CI 2-sided [0.022 to 0.120], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.073, 95% CI 2-sided [0.024 to 0.122], Standard Error of Mean 0.025 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9369, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.002, 95% CI 2-sided [-0.051 to 0.047], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

18. Secondary Outcome: Trough FVC Response on Day 43.
Description: as for outcome 17
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 43
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.150 (0.018) | 0.206 (0.018) | 0.213 (0.018) | 0.254 (0.018) | 0.318 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.168, 95% CI 2-sided [0.119 to 0.217], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.105, 95% CI 2-sided [0.056 to 0.154], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.103, 95% CI 2-sided [0.054 to 0.152], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0585, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.047, 95% CI 2-sided [-0.002 to 0.096], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.1042, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.041, 95% CI 2-sided [-0.008 to 0.090], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0097, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.065, 95% CI 2-sided [0.016 to 0.114], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.112, 95% CI 2-sided [0.063 to 0.161], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0120, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.063, 95% CI 2-sided [0.014 to 0.112], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0250, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.056, 95% CI 2-sided [0.007 to 0.105], Standard Error of Mean 0.025 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7889, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.007, 95% CI 2-sided [-0.042 to 0.056], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

19. Secondary Outcome: Trough FVC Response on Day 85.
Description: as for outcome 17
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and on day 85
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.077 (0.018) | 0.168 (0.018) | 0.144 (0.018) | 0.230 (0.018) | 0.265 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.187, 95% CI 2-sided [0.138 to 0.237], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.121, 95% CI 2-sided [0.072 to 0.170], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.153, 95% CI 2-sided [0.103 to 0.202], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0134, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.062, 95% CI 2-sided [0.013 to 0.111], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.086, 95% CI 2-sided [0.037 to 0.136], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1670, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.035, 95% CI 2-sided [-0.015 to 0.084], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.097, 95% CI 2-sided [0.048 to 0.146], Standard Error of Mean 0.025 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0085, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.066, 95% CI 2-sided [0.017 to 0.115], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.090, 95% CI 2-sided [0.041 to 0.140], Standard Error of Mean 0.025 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.3332, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.024, 95% CI 2-sided [-0.074 to 0.025], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

20. Secondary Outcome: Trough FVC Response on Day 170.
Description: Trough FVC was defined as the FVC value at the end of the dosing interval (24 hours) and was calculated as the mean of the 2 FVC measurements performed at 23h and at 23h 50 min after inhalation of study medication at the clinic visit on the previous day.
  Trough FVC response was defined as trough FVC minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an MMRM including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.093 (0.017) | 0.184 (0.017) | 0.169 (0.017) | 0.225 (0.017) | 0.246 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.153, 95% CI 2-sided [0.105 to 0.201], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.077, 95% CI 2-sided [0.029 to 0.125], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.132, 95% CI 2-sided [0.084 to 0.180], Standard Error of Mean 0.025 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0926, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.041, 95% CI 2-sided [-0.007 to 0.089], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0231, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.055, 95% CI 2-sided [0.008 to 0.103], Standard Error of Mean 0.024 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.3802, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.021, 95% CI 2-sided [-0.026 to 0.069], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0105, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.062, 95% CI 2-sided [0.015 to 0.110], Standard Error of Mean 0.024 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.076, 95% CI 2-sided [0.028 to 0.125], Standard Error of Mean 0.025 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.091, 95% CI 2-sided [0.043 to 0.139], Standard Error of Mean 0.025 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.5554, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.014, 95% CI 2-sided [-0.062 to 0.034], Standard Error of Mean 0.024 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

21. Secondary Outcome: Trough FVC Response on Day 365.
Description: as for outcome 17
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and on Day 365.
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 519 | 519 | 520 | 518 | 521
Litres | 0.014 (0.018) | 0.114 (0.018) | 0.108 (0.018) | 0.155 (0.018) | 0.191 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.178, 95% CI 2-sided [0.127 to 0.228], Standard Error of Mean 0.026 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.084, 95% CI 2-sided [0.033 to 0.134], Standard Error of Mean 0.026 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.142, 95% CI 2-sided [0.091 to 0.192], Standard Error of Mean 0.026 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.1112, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.041, 95% CI 2-sided [-0.009 to 0.091], Standard Error of Mean 0.026 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0632, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.048, 95% CI 2-sided [-0.003 to 0.098], Standard Error of Mean 0.026 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1615, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.036, 95% CI 2-sided [-0.014 to 0.086], Standard Error of Mean 0.026 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0027, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.077, 95% CI 2-sided [0.027 to 0.127], Standard Error of Mean 0.026 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.094, 95% CI 2-sided [0.044 to 0.144], Standard Error of Mean 0.026 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.101, 95% CI 2-sided [0.050 to 0.151], Standard Error of Mean 0.026 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7925, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.007, 95% CI 2-sided [-0.057 to 0.044], Standard Error of Mean 0.026 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

22. Secondary Outcome: FEV1 AUC(0-12h) Response in the Sub-set of Patients With 12-hour Pulmonary Function Test (PFT) on Day 169 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: FEV1 AUC(0-12h) was calculated as the area under the FEV1- time curve from 0 to 12 h post-dose using the trapezoidal rule, divided by the duration (12 h) to report in litres.
  FEV1 AUC(0-12h) response was defined as FEV1 AUC(0-12h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate.
  Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 169 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h post-dose on Day 169.
Population: 12 hr PFT set: All patients who have given Informed Consent for the 12-hour PFT testing and had any spirometry measurement after 3-hour and before or at 12-hours post-dose on Days 169 and 170.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.131 (0.015) | 0.109 (0.016) | 0.127 (0.017) | 0.202 (0.016) | 0.250 (0.016)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.118, 95% CI 2-sided [0.074 to 0.162], Standard Error of Mean 0.022 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.123, 95% CI 2-sided [0.077 to 0.169], Standard Error of Mean 0.023 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg)
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0012, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.071, 95% CI 2-sided [0.028 to 0.114], Standard Error of Mean 0.022 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.094, 95% CI 2-sided [0.050 to 0.137], Standard Error of Mean 0.022 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg)
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0010, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.076, 95% CI 2-sided [0.031 to 0.121], Standard Error of Mean 0.023 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg)
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0384, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.047, 95% CI 2-sided [0.003 to 0.092], Standard Error of Mean 0.023 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg)
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.141, 95% CI 2-sided [0.097 to 0.185], Standard Error of Mean 0.022 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg)
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8428, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.004, 95% CI 2-sided [-0.049 to 0.040], Standard Error of Mean 0.023 — Tiotropium (5 µg) versus Olodaterol (5 µg)
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.3048, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.022, 95% CI 2-sided [-0.065 to 0.020], Standard Error of Mean 0.022 — Tiotropium (2.5 µg) versus Olodaterol (5 µg)
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4311, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.018, 95% CI 2-sided [-0.027 to 0.063], Standard Error of Mean 0.023 — Tiotropium (5 µg) versus Tiotropium (2.5 µg)

23. Secondary Outcome: FEV1 AUC(0-24h) Response in the Sub-set of Patients With 12-h PFTs on Day 169 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: FEV1 AUC(0-24h) was calculated as the area under the FEV1- time curve from 0 to 24 h post-dose using the trapezoidal rule, divided by the duration (24 h) to report in litres. FEV1 AUC(0-24h) response was defined as FEV1 AUC(0-24h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate.
  Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 169 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 23 h, 23 h and 50 min post-dose on Day 169.
Population: 12-hr PFT set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.108 (0.014) | 0.083 (0.015) | 0.100 (0.016) | 0.159 (0.015) | 0.206 (0.015)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.098, 95% CI 2-sided [0.057 to 0.139], Standard Error of Mean 0.021 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.106, 95% CI 2-sided [0.063 to 0.149], Standard Error of Mean 0.022 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg)
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0136, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.051, 95% CI 2-sided [0.010 to 0.091], Standard Error of Mean 0.021 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0003, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.075, 95% CI 2-sided [0.035 to 0.116], Standard Error of Mean 0.021 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg)
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0065, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.059, 95% CI 2-sided [0.016 to 0.101], Standard Error of Mean 0.022 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg)
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0277, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.047, 95% CI 2-sided [0.005 to 0.089], Standard Error of Mean 0.021 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg)
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.122, 95% CI 2-sided [0.081 to 0.164], Standard Error of Mean 0.021 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg)
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7116, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.008, 95% CI 2-sided [-0.049 to 0.034], Standard Error of Mean 0.021 — Tiotropium (5 µg) versus Olodaterol (5 µg)
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2332, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.024, 95% CI 2-sided [-0.065 to 0.016], Standard Error of Mean 0.020 — Tiotropium (2.5 µg) versus Olodaterol (5 µg)
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4374, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.017, 95% CI 2-sided [-0.025 to 0.059], Standard Error of Mean 0.021 — Tiotropium (5 µg) versus Tiotropium (2.5 µg)

24. Secondary Outcome: FVC AUC(0-12h) Response in the Sub-set of Patients With 12-h PFTs on Day 169 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: FVC AUC(0-12h) was calculated as the area under the FVC- time curve from 0 to 12 h post-dose using the trapezoidal rule, divided by the duration (12 h) to report in litres.
  FVC AUC(0-12h) response was defined as FVC AUC(0-12h) minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate. Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: as for outcome 22
Population: 12-hr PFT set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.227 (0.029) | 0.180 (0.030) | 0.248 (0.032) | 0.356 (0.030) | 0.388 (0.031)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0002, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.161, 95% CI 2-sided [0.077 to 0.244], Standard Error of Mean 0.043 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0017, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.140, 95% CI 2-sided [0.053 to 0.228], Standard Error of Mean 0.045 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg)
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0022, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.128, 95% CI 2-sided [0.046 to 0.210], Standard Error of Mean 0.042 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.176, 95% CI 2-sided [0.093 to 0.259], Standard Error of Mean 0.042 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg)
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0141, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.108, 95% CI 2-sided [0.022 to 0.194], Standard Error of Mean 0.044 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg)
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4581, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.032, 95% CI 2-sided [-0.053 to 0.118], Standard Error of Mean 0.043 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg)
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.208, 95% CI 2-sided [0.124 to 0.293], Standard Error of Mean 0.043 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg)
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6335, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.021, 95% CI 2-sided [-0.064 to 0.105], Standard Error of Mean 0.043 — Tiotropium (5 µg) versus Olodaterol (5 µg)
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2530, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.047, 95% CI 2-sided [-0.129 to 0.034], Standard Error of Mean 0.041 — Tiotropium (2.5 µg) versus Olodaterol (5 µg)
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1188, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.068, 95% CI 2-sided [-0.017 to 0.153], Standard Error of Mean 0.043 — Tiotropium (5 µg) versus Tiotropium (2.5 µg)

25. Secondary Outcome: FVC AUC(0-24h) Response in Sub-set of Patients With 24-h PFTs on Day 169 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: FVC AUC(0-24h) was calculated as the area under the FVC- time curve from 0 to 24 h post-dose using the trapezoidal rule, divided by the duration (24 h) to report in litres.
  FVC AUC(0-24h) response was defined as FVC AUC(0-24h) minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate.
  Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: as for outcome 23
Population: 12-hr PFT set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.192 (0.028) | 0.141 (0.028) | 0.203 (0.030) | 0.297 (0.029) | 0.329 (0.030)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0008, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.137, 95% CI 2-sided [0.057 to 0.217], Standard Error of Mean 0.041 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0032, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.126, 95% CI 2-sided [0.042 to 0.209], Standard Error of Mean 0.043 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg)
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0085, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.105, 95% CI 2-sided [0.027 to 0.183], Standard Error of Mean 0.040 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg)
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.156, 95% CI 2-sided [0.077 to 0.235], Standard Error of Mean 0.040 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg)
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0255, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.094, 95% CI 2-sided [0.011 to 0.176], Standard Error of Mean 0.042 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg)
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4393, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.032, 95% CI 2-sided [-0.049 to 0.113], Standard Error of Mean 0.041 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg)
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.188, 95% CI 2-sided [0.108 to 0.269], Standard Error of Mean 0.041 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg)
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7784, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.012, 95% CI 2-sided [-0.069 to 0.092], Standard Error of Mean 0.041 — Tiotropium (5 µg) versus Olodaterol (5 µg)
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1965, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.051, 95% CI 2-sided [-0.129 to 0.026], Standard Error of Mean 0.039 — Tiotropium (2.5 µg) versus Olodaterol (5 µg)
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1315, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.063, 95% CI 2-sided [-0.019 to 0.144], Standard Error of Mean 0.041 — Tiotropium (5 µg) versus Tiotropium (2.5 µg)

26. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score on Day 85 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: as for outcome 3
Time Frame: Day 85
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 954 | 960 | 955 | 990 | 979
points on a scale | 38.832 (0.398) | 37.821 (0.397) | 37.822 (0.399) | 37.304 (0.392) | 36.691 (0.394)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -2.141, 95% CI 2-sided [-3.239 to -1.043], Standard Error of Mean 0.560 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0435, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.131, 95% CI 2-sided [-2.230 to -0.033], Standard Error of Mean 0.560 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg)
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0063, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.528, 95% CI 2-sided [-2.623 to -0.432], Standard Error of Mean 0.559 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.3545, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.517, 95% CI 2-sided [-1.611 to 0.577], Standard Error of Mean 0.558 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.3542, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.518, 95% CI 2-sided [-1.614 to 0.578], Standard Error of Mean 0.559 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2697, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.613, 95% CI 2-sided [-1.702 to 0.476], Standard Error of Mean 0.556 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0434, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.130, 95% CI 2-sided [-2.227 to -0.033], Standard Error of Mean 0.559 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0732, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.010, 95% CI 2-sided [-2.114 to 0.095], Standard Error of Mean 0.563 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0724, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.011, 95% CI 2-sided [-2.114 to 0.092], Standard Error of Mean 0.563 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9983, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.001, 95% CI 2-sided [-1.102 to 1.104], Standard Error of Mean 0.563 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

27. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score on Day 365 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: as for outcome 3
Time Frame: Day 365
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 954 | 960 | 955 | 990 | 979
points on a scale | 38.989 (0.414) | 37.609 (0.409) | 37.581 (0.411) | 37.553 (0.403) | 37.138 (0.404)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.852, 95% CI 2-sided [-2.985 to -0.718], Standard Error of Mean 0.578 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4413, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.444, 95% CI 2-sided [-1.573 to 0.686], Standard Error of Mean 0.576 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.437, 95% CI 2-sided [-2.569 to -0.304], Standard Error of Mean 0.578 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.9222, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.056, 95% CI 2-sided [-1.182 to 1.070], Standard Error of Mean 0.574 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.9602, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.029, 95% CI 2-sided [-1.157 to 1.100], Standard Error of Mean 0.576 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4669, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.415, 95% CI 2-sided [-1.533 to 0.703], Standard Error of Mean 0.570 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4126, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.471, 95% CI 2-sided [-1.598 to 0.656], Standard Error of Mean 0.575 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0158, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.408, 95% CI 2-sided [-2.551 to -0.265], Standard Error of Mean 0.583 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0177, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.381, 95% CI 2-sided [-2.521 to -0.240], Standard Error of Mean 0.582 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9624, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.027, 95% CI 2-sided [-1.164 to 1.109], Standard Error of Mean 0.580 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

28. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 43 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: Mahler Transitional Dyspnoea Index (TDI) focal score on Day 43 From the Two Twin Trials, present 1237.5 (NCT01431274) and 1237.6 (NCT01431287).
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome. Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 43
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.453 (0.096) | 1.430 (0.097) | 1.408 (0.097) | 1.876 (0.096) | 2.048 (0.096)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.595, 95% CI 2-sided [0.329 to 0.862], Standard Error of Mean 0.136 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.640, 95% CI 2-sided [0.373 to 0.907], Standard Error of Mean 0.136 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.423, 95% CI 2-sided [0.156 to 0.690], Standard Error of Mean 0.136 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.446, 95% CI 2-sided [0.179 to 0.712], Standard Error of Mean 0.136 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.468, 95% CI 2-sided [0.201 to 0.735], Standard Error of Mean 0.136 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2045, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.172, 95% CI 2-sided [-0.094 to 0.438], Standard Error of Mean 0.136 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.618, 95% CI 2-sided [0.351 to 0.885], Standard Error of Mean 0.136 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7432, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.045, 95% CI 2-sided [-0.313 to 0.223], Standard Error of Mean 0.137 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.8687, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.023, 95% CI 2-sided [-0.290 to 0.245], Standard Error of Mean 0.136 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8709, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.022, 95% CI 2-sided [-0.290 to 0.246], Standard Error of Mean 0.137 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

29. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 85 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: Mahler Transitional Dyspnoea Index (TDI) focal score on Day 85 From the Two Twin Trials, present 1237.5 (NCT01431274) and 1237.6 (NCT01431287).
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 85
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.506 (0.097) | 1.698 (0.097) | 1.702 (0.097) | 1.925 (0.096) | 2.136 (0.096)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.630, 95% CI 2-sided [0.362 to 0.898], Standard Error of Mean 0.137 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.434, 95% CI 2-sided [0.166 to 0.703], Standard Error of Mean 0.137 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.419, 95% CI 2-sided [0.151 to 0.687], Standard Error of Mean 0.137 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0966, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.227, 95% CI 2-sided [-0.041 to 0.495], Standard Error of Mean 0.137 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.1029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.223, 95% CI 2-sided [-0.045 to 0.492], Standard Error of Mean 0.137 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1220, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.211, 95% CI 2-sided [-0.056 to 0.478], Standard Error of Mean 0.136 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.438, 95% CI 2-sided [0.170 to 0.707], Standard Error of Mean 0.137 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1542, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.196, 95% CI 2-sided [-0.074 to 0.465], Standard Error of Mean 0.137 — Tiotropium (5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1626, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.192, 95% CI 2-sided [-0.077 to 0.461], Standard Error of Mean 0.137 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9765, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.004, 95% CI 2-sided [-0.265 to 0.274], Standard Error of Mean 0.138 — Tiotropium (5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors

30. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 365 From the Two Twin Trials, Present 1237.5 (NCT01431274) and 1237.6 (NCT01431287)
Description: Mahler Transitional Dyspnoea Index (TDI) focal score on Day 365 From the Two Twin Trials, present 1237.5 (NCT01431274) and 1237.6 (NCT01431287).
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome. Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 365
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.411 (0.101) | 1.450 (0.100) | 1.736 (0.101) | 1.782 (0.099) | 2.058 (0.099)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.647, 95% CI 2-sided [0.370 to 0.925], Standard Error of Mean 0.142 — Tio+Olo FDC (5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0226, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.322, 95% CI 2-sided [0.045 to 0.600], Standard Error of Mean 0.141 — Tio+Olo FDC (5/5 μg) versus Tiotropium (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.371, 95% CI 2-sided [0.093 to 0.649], Standard Error of Mean 0.142 — Tio+Olo FDC (2.5/5 μg) versus Olodaterol (5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0186, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.332, 95% CI 2-sided [0.056 to 0.609], Standard Error of Mean 0.141 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.7441, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.046, 95% CI 2-sided [-0.231 to 0.324], Standard Error of Mean 0.142 — Tio+Olo FDC (2.5/5 μg) versus Tiotropium (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0492, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.276, 95% CI 2-sided [0.001 to 0.551], Standard Error of Mean 0.140 — Tio+Olo FDC (5/5 µg) versus Tio+Olo FDC (2.5/5 μg). Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.608, 95% CI 2-sided [0.332 to 0.884], Standard Error of Mean 0.141 — Tio+Olo FDC (5/5 µg) versus Tiotropium (2.5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0230, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.325, 95% CI 2-sided [0.045 to 0.605], Standard Error of Mean 0.143 — Tiotropium (2.5 µg) versus Olodaterol (5 µg) Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.7855, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.039, 95% CI 2-sided [-0.240 to 0.317], Standard Error of Mean 0.142 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0442, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.286, 95% CI 2-sided [0.007 to 0.564], Standard Error of Mean 0.142 — Tiotropium (2.5 µg) versus Olodaterol (5 µg). Spatial power covariance structure for within-patient errors

ADVERSE EVENTS:
Time Frame: All Adverse events with an onset after the first dose of study medication up to a period of 21 days after the last dose of study medication were assigned to the treatment period for evaluation (Up to 447 days)
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Serious Adverse Events (participants affected / at risk) | 75/528 | 66/525 | 79/527 | 81/522 | 87/522
Other Adverse Events (participants affected / at risk) | 221/528 | 207/525 | 210/527 | 211/522 | 193/522
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5 μg) (N=528) | Tiotropium (2.5 μg) (N=525) | Tiotropium (5 μg) (N=527) | Tio+Olo FDC (2.5/5 μg) (N=522) | Tio+Olo FDC (5/5 μg) (N=522)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 0 | 4
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 2 | 2 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 1 | 1
Electrocution (General disorders) | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0 | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infected bites (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 3 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 8 | 5 | 5 | 10 | 9
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Arteriogram coronary (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Fascial hernia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Enchondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 5 | 3 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 2 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Critical illness polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 2 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 1 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 | 25 | 24 | 20 | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Nasal septal operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5 μg) (N=528) | Tiotropium (2.5 μg) (N=525) | Tiotropium (5 μg) (N=527) | Tio+Olo FDC (2.5/5 μg) (N=522) | Tio+Olo FDC (5/5 μg) (N=522)
Nasopharyngitis (Infections and infestations) | 65 | 64 | 67 | 64 | 67
Upper respiratory tract infection (Infections and infestations) | 24 | 30 | 30 | 40 | 25
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 155 | 144 | 151 | 133 | 134

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.